CLINICAL TRIAL: NCT06251544
Title: (TRAILBLASER) TRAIL-R2 and HER2 Bi-Specific Chimeric Antigen Receptor T Cells for the Treatment of Metastatic Breast Cancer
Brief Title: TRAIL-R2 and HER2 Bi-Specific Chimeric Antigen Receptor (CAR) T Cells for the Treatment of Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Valentina Hoyos, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-54673 TRAILBLASER
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Tumor, Breast; Breast Tumor; Malignant Neoplasm of Breast; Mammary Cancer; Mammary Neoplasm; Mammary Neoplasms, Human; Neoplasm, Breast
Keywords: HER2 positive
MeSH Terms: conditions — Breast Neoplasms; Mammary Neoplasms, Animal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: HTR2 T Cells (without lymphodepletion) (Experimental): Two dose levels will be evaluated in Arm A (without lymphodepletion)
  Interventions: Genetic: HTR2 T Cells
- Arm B: HTR2 T Cells (with lymphodepletion) (Experimental): Two dose levels will be evaluated in Arm B (with lymphodepletion)
  Interventions: Genetic: HTR2 T Cells

INTERVENTIONS:
Genetic: HTR2 T Cells — Arm A -- Two dose levels will be evaluated:
  Dose level One: 1.00E+06
  Dose level Two: 1.00E+07
  Arms: Arm A: HTR2 T Cells (without lymphodepletion)
Genetic: HTR2 T Cells — Arm B -- Two dose levels will be evaluated:
  Dose level Two: 1.00E+07
  Dose Level Three: 1.00E+08
  Arms: Arm B: HTR2 T Cells (with lymphodepletion)

SUMMARY:
The purpose of this study is to find the biggest dose of HTR2 T cells that is safe, to see how long these cells last in the body, to learn the side effects, and to see if these cells are able to fight and kill HER2 expressing breast cancer.

Patients eligible for this study have metastatic breast cancer that has HER2 expression and has progressed on at least one line of therapy. This is a gene transfer research study using special immune cells called T cells. T cells are a type of white blood cell that helps the body recognize and fight cancer cells.

The body has different ways of fighting diseases and no single way seems perfect for fighting cancer. This research combines two different ways of fighting cancer: antibodies and T cells. Antibodies are proteins that protect the body from infectious disease and possibly cancer. T cells, or T lymphocytes, are special blood cells that can kill other cells, including tumor cells. Both antibodies and T cells have shown promise treating cancer but have not been strong enough to cure most patients.

Previous research has found that investigators can put genes into T cells that helps them recognize cancer cells and kill them. Investigators now want to see if by putting a new gene in those T cells to help recognize breast cancer cells expressing HER2 can kill the cancer cells. In clinical trials for various cancer types that express HER2, our center engineered a CAR that recognizes HER2 and put this CAR into patients own T cells and gave them back. Investigators saw that the cells did grow and patients did tolerate and respond to the treatment.

Investigators will add a gene to the HER2 recognizing CAR T cells that will improve the T cells function. Investigators know that some immune cells in the body can lower T cells ability to kill cancer cells. Investigators have identified an antibody that will inactivate those immune suppressive cells thereby allowing T cells to survive better to recognize and kill cancer cells. This antibody targets the Trail-R2 receptor and is referred to as TR2.

Also, investigators know that T cells need the support of cytokines to perform their immune functions. There is evidence showing that the addition of interleukin 15 (IL15) enhances CAR T cells ability to kill cancer cells. As a result, investigators also added IL15 to the HER2 and TR2 targeting CAR T cells (HTR2 T cells).

The HTR2 T cells are an investigational product not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
To make the T cells, the investigators will take the patient's blood and stimulate it with growth factors to make T cells grow. Investigators use a retrovirus to insert HER CAR, TR2 antibody and IL 15 genes into the T cells.

HTR2 cells are generated from the patient's T cells and are frozen. At the time the patient is scheduled to be treated, the cells will then be thawed and injected into the patient over 5 to 10 minutes. Patients will only get one dose of HTR2 T cells during the infusion. If the patient has a good response and tolerance, we may be able to repeat infusion in the future. The patent may be pretreated with Tylenol and Benadryl to prevent possible allergic reaction to the T cell administration.

If investigators need to stop the HTR2 T cells due to bad side effects, investigators have inserted a gene called iCasp9 into the T cells. This allows investigators to eliminate the HTR2 T cells in the blood when the gene comes into contact with a medication called Rimiducid. The drug Rimiducid is not yet FDA approved and is an experimental drug, but it has been tested in humans without bad side-effects. Investigators will only use this drug to kill the T cells if necessary due to side effects. Since investigators do not know exactly what dose will effectively stop HTR2 T cells in individual patients, investigators will start at a low dose with the ability to increase the dose two more times based on how patients are doing. Blood work will be done to ensure that the HTR2 T cells have been successfully eliminated.

The treatment will be given by the Center for Cell and Gene Therapy at Houston Methodist Hospital.

MEDICAL TESTS BEFORE TREATMENT

Before being treated, patients will receive a series of standard medical tests:

* Physical exam and history
* Blood tests to measure blood cells and organ function
* Measurements of the tumor by scans at baseline prior to treatment
* Ultrasound of the heart to make sure the patient has good baseline cardiac function

Additionally, patients will need a biopsy of their tumor tissue to both confirm HER2 expression and to be used for research purposes.

MEDICAL TESTS DURING AND AFTER TREATMENT

Within four weeks after infusion, patients will be monitored on a weekly basis for dose limiting side effects of the HTR2 T cells:

* Physical exam and history
* Blood tests to measure blood cells and organ function

After the initial six weeks, patients will be monitored at a minimum every 3 months for the 1st year and every 6 months between 1 to year 5 or as frequently as deemed necessary:

* Physical exam and history
* Blood tests to measure blood cells and organ function
* Measurements of patient's tumor by scans to assess treatment response

To learn more about the way T cells work in the patient's body, investigators will obtain up to 50 ml of blood from patient before chemotherapy, before the T-cell infusion, 1 to 4 hours, 1, 2, 3, 4 weeks and 8 weeks after infusion, every 3 months for a year followed by every 6 months for 4 years and then every year for the the next 10 years. Total participation on this study will be 15 years. During the time points listed above, if the T cells are found in the blood at a certain amount, an extra half a tablespoon of blood may be needed for additional testing.

Investigators will obtain one tissue biopsy within 4 weeks after infusion and as clinically indicated thereafter. If additional clinically indicated tumor biopsies are obtained, investigators will ask for a portion of the sample for research.

ELIGIBILITY:
Procurement Inclusion Criteria:

1. Any patient between 18-80 years of age regardless of sex, with a diagnosis of metastatic or locally recurrent unresectable HER2 positive breast cancer.
2. HER2 tumor expression1+, 2+ or 3+ by IHC
3. The disease must have progressed after standard first line therapy. Patients are still eligible if they have failed more than one line of therapy.
4. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Treatment Inclusion Criteria:

1. Patients between ages 18 and 80 years old with a diagnosis of either stage IV breast cancer or locally recurrent unresectable breast cancer. Disease must have progressed after standard first line therapy. Patients are still eligible if they have failed more than one line of therapy.
2. Measurable or evaluable disease per RECIST 1.1 criteria.
3. HER2 tumor expression 1+, 2+ or 3+ by IHC.
4. Bilirubin ≤ 3x upper limit of normal.
5. AST and ALT ≤ 3x upper limit of normal
6. Hemoglobin ≥ 7 g/dl (may be transfused values)
7. Serum creatinine < 2 x the upper limit of normal.
8. Pulse oximetry of > 90% on room air.
9. Off conventional or investigational therapy for 3 weeks prior to study entry.
10. ECOG Performance Status ≤ 2
11. The patient is able to understand and give informed consent to study related procedures and treatments.

Procurement Exclusion Criteria:

1. Known pregnancy or actively breast feeding.
2. Active and uncontrolled bacterial, viral, or fungal infection.
3. Patients with current use of systemic corticosteroids (Prednisone equivalent >0.5mg/kg/day).
4. Patients with abnormal left ventricular function (LVEF <55%)
5. Patients with brain metastases that are progressing.

Treatment Exclusion Criteria:

1. Pregnant or breast feeding
2. Active and uncontrolled bacterial, viral or fungal infection
3. Patient with current use of systemic corticosteroids (prednisone equivalent >0.5 mg/kg/day.
4. Patients with abnormal left ventricular function (LVEF <55%).
5. Patients with brain metastases that are progressing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate | 4 weeks after first infusion
  Rate of incidents of dose limiting toxicity by dose levels.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3 months after first infusion
  Proportion of subjects with best overall response of complete response (CR) or partial response (PR) according to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Hoyos, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States